CLINICAL TRIAL: NCT04777253
Title: Effectiveness of Biofeedback Methods in Rehabilitation of Arm Function in Patients After Stroke
Brief Title: Rehabilitation of Arm Function Using a Biofeedback Method After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bogumiła Pniak (Other)
Responsible Party: Sponsor-Investigator, Bogumiła Pniak, MSc, University of Rzeszow
Organization: University of Rzeszow (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: stroke - biofeedback
Record Dates: First submitted 2021-02-11; First posted 2021-03-02 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Rehabilitation; Stroke; Biofeedback
Keywords: Health-resort based rehabilitation; Stroke; Biofeedback; Conventional (traditional) rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: random selection to two groups (study group and control group)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback method and Health-resort based rehabilitation (Experimental): Health-resort based treatments supplemented with biofeedback training
  Interventions: Other: Biofeedback method; Other: Health-resort based rehabilitation
- Health-resort based rehabilitation (Other): Control group - health-resort based treatments, without biofeedback training.
  Interventions: Other: Health-resort based rehabilitation

INTERVENTIONS:
Other: Biofeedback method — Patients in the study group will participate in training with visual biofeedback, aimed to improve motor function of the arm. The exercise will be performed using a Biometrics device. The biofeedback training will be carried out for 30 minutes per day.
  Health-resort based rehabilitation The patients will participate in a three-week rehabilitation program (from Monday to Friday), with the treatments and therapies continued for up to two hours per day.
  The program will include: group and individual exercise (active and assisted exercises, manipulation exercise, PNF-based practice, balance and breathing exercise), manual massage, physical treatments, such as: laser, whirlpool therapy, mud compress therapy, carbonic acid therapy, TENS therapy, BIO-V lamp, and localized cryotherapy.
  Arms: Biofeedback method and Health-resort based rehabilitation
Other: Health-resort based rehabilitation — The patients will participate in a three-week rehabilitation program (from Monday to Friday), with the treatments and therapies continued for up to two hours per day.
  The program will include: group and individual exercise (active and assisted exercises, manipulation exercise, PNF-based practice, balance and breathing exercise), manual massage, physical treatments, such as: laser, whirlpool therapy, mud compress therapy, carbonic acid therapy, TENS therapy, BIO-V lamp, and localized cryotherapy

SUMMARY:
The research will make it possible to assess effects of rehabilitation of arm function with the use of biofeedback method and conventional therapies administered to patients at a chronic stage of recovery post-stroke, as part of the treatment in a health-resort setting.

DETAILED DESCRIPTION:
: In accordance with the study design, the group will comprise 100 patients with hemiparesis after stroke, participating in a health-resort based rehabilitation program during their stay in the Health-Resort Rehabilitation Hospital in Iwonicz Zdrój, Poland. The minimum size of the sample was calculated based on the total annual number of patients after stroke receiving treatment in the Health-Resort Rehabilitation Hospital in Iwonicz Zdrój, i.e. approximately 200 patients, 100% of these being in a chronic stage of recovery. It was assumed that 50% of the patients would present stage 4-5 arm paresis according Brunnström scale. A fraction of 0.8 and a maximum error of 5% were applied and the sample size of 71 patients was obtained.

The patients meeting eligibility criteria will be randomly divided into two groups:

* the study group (50 patients), participating in a conventional rehabilitation program supplemented with additional biofeedback training;
* the control group (50 patients), participating in the conventional rehabilitation program only.

The patients in both groups will participate in a three-week rehabilitation program (from Monday to Friday), with the treatments and therapies continued for up to two hours per day. The program will include: group and individual exercise (active and assisted exercises, manipulation exercises, PNF-based practice, balance and breathing exercises), manual massage, physical treatments, such as: laser, whirlpool therapy, mud compress therapy, carbonic acid therapy, TENS therapy, BIO-V lamp, and localized cryotherapy. The patients in the study group will also receive biofeedback training aimed to improve motor function of the upper limb. The exercise will be performed using equipment manufactured by Biometrics. The device makes it possible to perform movements in all the planes of the joints in the upper limb. During the exercise, a visualisation of the movements is shown to the patient on the screen; this biofeedback makes it possible for them to regulate and increase the range of movement, to use greater muscle strength and to visually assess the accuracy of their performance. The training with the biofeedback function will be carried out for 30 minutes per day.

After the program is completed, the subjects from the control group will have an opportunity to also practice with the Biometrics device with the biofeedback function.

Examinations will be carried out three times: the baseline at the start of the rehabilitation program, a check-up at the end of the three-week program, and a follow-up two months after discharge from the hospital. The tests will be performed at the same time of day, and following the same conditions.

The patients' condition and the rehabilitation effects will be assessed using the following measures:

* hand grip strength and pinching strength of the fingers, to be tested with a dynamometer and pinch meter, respectively;
* ranges of motion in the joints of the upper limb, with R500 goniometer;
* manual skills, with Box and Blocks test;
* handgrip function, according Franchay scale;
* motor capacities of the upper limb, according to Fugl-Meyer Motor Assessment Scale;
* EMG test, with the Biometrics device;
* activities of daily living, with Barthel Index.

ELIGIBILITY:
Inclusion Criteria:

* informed, voluntary consent of the patient;
* a single ischemic stroke experienced;
* hemiparesis;
* a minimum of 6 months from the stroke onset;
* age 45-75 years;
* elementary (basic) handgrip ability;
* stage 4-5 arm paresis according Brunnström scale;
* stage 3 disability according to Rankin scale;
* spasticity in the paretic arm up to 1 plus on the modified Ashworth scale;
* current health status, confirmed by a medical examination, allowing the person to take part in the study and in the exercise.

Exclusion Criteria:

* lack of informed and voluntary consent of the patient;
* two or more strokes experienced, haemorrhagic stroke, brain stem and cerebellar stroke;
* impairments in higher mental functions adversely affecting the ability to understand and perform the tasks during exercise;
* visual field impairment;
* mechanical and thermal injuries potentially limiting handgrip function;
* coexisting neurological, rheumatic and orthopaedic conditions, including fixed contractures potentially affecting gripping abilities;
* unstable health condition;
* failure to complete the three-week rehabilitation program.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | : First examination - before the start of the rehabilitation program;
  measurements to be performed with a dynamometer The dynamometer registers strength lower than up to 90 kg,
Hand grip strength | Second examination - at the end of the three-week program
  measurements to be performed with a dynamometer The dynamometer registers strength lower than up to 90 kg,
Hand grip strength | Third examination - two months after discharge from the hospital (follow- up)
  measurements to be performed with a dynamometer The dynamometer registers strength lower than up to 90 kg,
pinching strength of the fingers | First examination - before the start of the rehabilitation program
  measurements to be performed with a pinch meter. The pinch meter registers strength lower than up to 22 kg.
pinching strength of the fingers | Second examination - at the end of the three-week program
  measurements to be performed with a pinch meter. The pinch meter registers strength lower than up to 22 kg.
pinching strength of the fingers | Third examination - two months after discharge from the hospital (follow- up)
  measurements to be performed with a pinch meter. The pinch meter registers strength lower than up to 22 kg.
Ranges of motion in the joints of the upper limb | First examination - before the start of the rehabilitation program
  with the use of R 500 goniometer; the device operates with an accuracy up to one degree.
Ranges of motion in the joints of the upper limb | Second examination - at the end of the three-week program
  with the use of R 500 goniometer; the device operates with an accuracy up to one degree.
Ranges of motion in the joints of the upper limb | Third examination - two months after discharge from the hospital (follow- up)
  with the use of R 500 goniometer; the device operates with an accuracy up to one degree.
EMG of extensors and flexors of the radiocarpal joint | First examination - before the start of the rehabilitation program
  EMG assessment of extensors and flexors of the radiocarpal joint on the Biometrics device
EMG of extensors and flexors of the radiocarpal joint | Second examination - at the end of the three-week program
  EMG assessment of extensors and flexors of the radiocarpal joint on the Biometrics device
EMG of extensors and flexors of the radiocarpal joint | Third examination - two months after discharge from the hospital (follow- up)
  EMG assessment of extensors and flexors of the radiocarpal joint on the Biometrics device

SECONDARY OUTCOMES:
Activities of daily living, assessed with Barthel Index. | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program; third examination - two months after discharge from the hospital (follow- up)
  Based on the scores assigned the patient's condition is described in the following way: I. 86-100 points - "slight" dependency; II. 21- 85 points - "moderately severe" dependency; III. 0 - 20 points - "severe" dependency.
  A maximum 100 points can be scored on Barthel scale.
Manual skills, assessed with Box and Blocks test; | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program; third examination - two months after discharge from the hospital (follow- up)
  The test uses a wooden box, divided into two equal parts by a partition, as well as 150 blocks. The subject moves as many blocks as possible from one part of the box to the other during 60 seconds.
Handgrip function, according Franchay scale | : First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program; third examination - two months after discharge from the hospital (follow- up)
  The scale consists of 7 tasks (pass/fail grading); the patient is awarded 1 point for each activity performed successfully, or 0 points for a failure to perform. The maximum score of seven points may be achieved for the performance of the tasks. Higher score corresponds to better manual skills. The scale measures the proximal control of the upper limb and the manual skills.
Motor capacities of the upper limb, according to Fugl-Meyer Motor Assessment Scale | First examination - before the start of the rehabilitation program; second examination - at the end of the three-week program; third examination - two months after discharge from the hospital (follow- up)
  Fugl-Meyer Motor Assessment Scale for Upper Extremity is a comprehensive tool enabling measurement of motor function; it comprises 33 motor tasks, designed to assess general movements, precision movements, grip, coordination and speed. It is also possible to perform H subgroup tests - assessing superficial and deep sensibility, and J subgroup tests - for range of passive motion and pain induced by such movements.
  Individual tasks are assessed on a scale 0-2 0 - impossible task
  1. - task partially completed,
  2. - task completed correctly The higher the score, the better.
Assessment of paretic limb function with the Brunnström scale. | Measurement during the patient's enrolment
  Motor performance (function) of extremities is to be assessed using Brunnström scale. This is a six-point scale designed to evaluate performance (function) of paretic extremities.The higher the score, the better.
  1-No moves 6-Precise movements, ball throw, button fastening and unfastening
Muscle tone (spasticity) will be examined with modified Ashworth scale. | Measurement during the patient's enrolment
  Increased muscle tone (spasticity) is to be examined with modified Ashworth scale. This is a six-point scale modified to include grade 1.
  0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM;
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moped;
  3. Considerable increase in muscle tone, passive movement difficult;
  4. Affected part(s) rigid in flexion or extension.
Assessment of disability level, using the modified Rankin scale (MRS) | : Measurement during the patient's enrolment
  Assessment of disability using the modified Rankin scale (MRS)
  Score Description 0 - No symptoms at all
  1- No significant disability despite symptoms; able to carry out all usual duties and activities; 2 - Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance; 3 - Moderate disability; requiring some help, but able to walk without assistance; 4 - Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance; 5 - Severe disability; bedridden, incontinent and requiring constant nursing care and attention; 6 - Dead TOTAL (0-6):

CONTACTS AND LOCATIONS:
Overall Officials: Bogumiła Pniak, MSc, Principal Investigator — University of Rzeszow
Locations (1):
- University of Rzeszów, Rzeszów, Poland